CLINICAL TRIAL: NCT03614637
Title: Cannabis Use and Epigenetic Alterations in Human Male Sperm Cells: Effects of Exposure and Abstinence (Component 1)
Brief Title: Cannabis Use and Epigenetic Alterations in Human Male Sperm Cells
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: John Templeton Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00086400
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-11

CONDITIONS: Cannabis Use
Keywords: Cannabis Abstinence Sperm Cells

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cannabis User Group: Forty eight participants who are regular Cannabis users with a self-reported frequency of at least once weekly over the past 6 months of screening visit.
  Interventions: Other: Cannabis use abstinence for 11 weeks
- Non-Cannabis User Group: Twenty four participants who self-report no Cannabis use in the past 6 months of screening visit and fewer than 10 times during their lifetime

INTERVENTIONS:
Other: Cannabis use abstinence for 11 weeks — Cannabis user group will be asked to abstain from any form of Cannabis use for 11 weeks. During their contingency management phase/abstinence phase, they will be required to come to the clinic for 25 visits over an 11 week period of abstinence.
  Groups: Cannabis User Group

SUMMARY:
This is a follow-up project to a proof-of-concept study to determine if Cannabis use in male humans is associated with changes in deoxyribonucleic acid (DNA) methylation profile of sperm. This proposal will examine the epigenome of sperm from men actively using Cannabis before and after a period of Cannabis abstinence. The results will be compared to control non-users.

DETAILED DESCRIPTION:
This project involves recruitment of 72 healthy males between the ages of 18 and 40 years. Forty eight of the participants will be regular cannabis users with a self-reported frequency of at least once weekly over the past 6 months, and a control group of twenty four cannabis non-users. Cannabis users will be asked to quit using cannabis for 11 weeks and will be required to attend 25 visits during the 11 week abstinence/contingency management period. Non-users will be asked to return to the clinic once a week for 11 weeks. Abstinence will be determined by self-report, qualitative urine rapid screening test at the clinic and quantitatively via Enzyme Immunoassay (EIA) analysis of THC (cannabinoids) and, by Liquid Chromatography Tandem Mass Spectrometry (LCMSMS) analysis of 11-nor-9-carboxy-∆ 9-tetrahydrocannabinol (THCCOOH) performed by an analytical lab contracted by the study team. Semen sample for both groups will be collected prior to the start of abstinence and after 11 weeks. Semen analysis and DNA methylation of sperm cells will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Between the ages of 18-40 years, inclusive;
* Free from significant medical/psychiatric conditions
* Willingness to provide baseline semen sample and again at the end of study participation
* Willingness to comply
* Ability to communicate verbally and in written form in English.

For the CANNABIS USER group:

* Self-reported Cannabis use of at least once weekly for past 6 months;
* THC level of at least 50 ng/ml (EIA, non-creatinine adjusted value) and THCCOOH level of at least 15ng/ml (LCMSMS, non-creatinine adjusted value);
* Positive result on urine rapid screening test for THC; and
* Willingness to abstain from Cannabis for 11 weeks during the course of the study

For the CANNABIS NON-USER group:

* Self-report of no Cannabis use in the past 6 months; fewer than 10 times lifetime;
* THCCOOH level = 0 ng/ml; (EIA non-creatinine adjusted value) and
* Negative result on urine rapid screening test.

Exclusion Criteria:

* Positive result for any other drugs of abuse on urine rapid screening test (including cocaine, methamphetamine, opiates, benzodiazepines, and barbiturates); or use of nicotine or tobacco products;-Currently prescribed any psychoactive medication;
* Current diagnosis of any significant psychiatric condition, including substance use disorders. For the user group, Cannabis Use Disorder that does not require immediate clinical attention in the opinion of the clinician/investigator will be allowed.
* Score on the Marijuana Screening Inventory-X > 10;
* Score on the Alcohol Use Disorders Identification Test > 8;
* Expired breath CO reading of > 8 ppm at screening and throughout the study.
* Expired Breath Alcohol Level of > 0.000 at screening.
* Urinary cotinine level greater than 2- indicating urinary concentrations of > 30ng/ml cotinine at screening and throughout the study
* Estimated IQ < 80 as assessed by the Kaufman Brief Intelligence Test, Second Edition; and
* Unable to comply with study requirements or otherwise unsuitable for participation in the opinion of the study physician and/or study psychologist.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We are looking at effects of Cannabis use in sperm cells.
Study Population: 72 healthy males between the ages of 18 and 40 years. Forty eight - regular Cannabis users with a self-reported frequency of at least once weekly over the past 6 months, Twenty four Cannabis non-users - control group
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Group differences in sperm DNA methylation profiles between user and non-user group | Baseline
  We will compare the overall DNA methylation profiles in sperm cells of user and non-user group to replicate findings in the pilot study.
Within group change in DNA methylation profiles from baseline to after 11 weeks of Cannabis abstinence | Baseline to after 11 weeks of abstinence from Cannabis use.
  We will compare the overall DNA methylation profiles in sperm cells after an 11 week period of Cannabis abstinence in the user group

SECONDARY OUTCOMES:
Group differences in the sperm analysis profile between user and non-user group | Baseline
  We will compare the overall sperm analysis profile of user versus non-user group to replicate findings in the pilot study
Within group change in sperm analysis profile from baseline to after eleven weeks of Cannabis abstinence | Baseline to after 11 weeks of abstinence from Cannabis use
  We will compare sperm analysis profile after an eleven week period of Cannabis abstinence in the user group

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States